CLINICAL TRIAL: NCT00335452
Title: Randomized, Multinational, Double-blind Study, Comparing a High Loading Dose Regimen of Clopidogrel Versus Standard Dose in Patients With Unstable Angina or Myocardial Infarction Managed With an Early Invasive Strategy.
Brief Title: Clopidogrel Optimal Loading Dose Usage to Reduce Recurrent EveNTs/Optimal Antiplatelet Strategy for InterventionS
Acronym: CURRENT/OASIS7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: ICD, sanofi-aventis
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5965; EUDRACT: 2006-000313-38
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Acute Coronary Disease; Angina Unstable
Keywords: platelet aggregation inhibitors; acute coronary disease; percutaneous coronary
MeSH Terms: conditions — Angina, Unstable | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clopidogrel high dose treatment regimen + ASA high dose (Experimental)
  Interventions: Drug: Clopidogrel; Drug: acetylsalicyclic acid (ASA)
- Clopidogrel high dose treatment regimen + ASA low dose (Experimental)
  Interventions: Drug: Clopidogrel; Drug: acetylsalicyclic acid (ASA)
- Clopidogrel standard treatment regimen + ASA high dose (Active Comparator)
  Interventions: Drug: Clopidogrel; Drug: acetylsalicyclic acid (ASA)
- Clopidogrel standard treatment regimen + ASA low dose (Active Comparator)
  Interventions: Drug: Clopidogrel; Drug: acetylsalicyclic acid (ASA)

INTERVENTIONS:
Drug: Clopidogrel — oral administration
  Other Names: SR25990; Plavix
Drug: acetylsalicyclic acid (ASA) — oral administration

SUMMARY:
The purpose of this study is to evaluate whether a higher dosage of clopidogrel with aspirin (two doses) will decrease the risk of ischemic complications (cardiac death (CV death), myocardial infarction (MI), stroke) after a percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute coronary disease with clinical symptoms and at least electrocardiogram changes or cardiac enzymes elevated

Exclusion Criteria:

* Use of anticoagulants within 10 days with an international normalized ratio (INR) > 1.5 or planned use during the hospitalisation period
* Administration of clopidogrel > 75 mg prior to randomization
* Contraindication to clopidogrel or aspirin
* Active bleeding or significant risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25086 (Actual)
Dates: Start 2006-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamir MEHTA, MD, Principal Investigator — Hamilton General Hospital, McMaster University, CANADA
Locations (38):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Beijing, China
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Riga, Latvia
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Admnistrative Office, Madrid, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom

REFERENCES:
- [Result] CURRENT-OASIS 7 Investigators; Mehta SR, Bassand JP, Chrolavicius S, Diaz R, Eikelboom JW, Fox KA, Granger CB, Jolly S, Joyner CD, Rupprecht HJ, Widimsky P, Afzal R, Pogue J, Yusuf S. Dose comparisons of clopidogrel and aspirin in acute coronary syndromes. N Engl J Med. 2010 Sep 2;363(10):930-42. doi: 10.1056/NEJMoa0909475. PMID 20818903
- [Result] Fuster V. Fine-tuning therapy for acute coronary syndromes. N Engl J Med. 2010 Sep 2;363(10):976-7. doi: 10.1056/NEJMe1008891. No abstract available. PMID 20818910
- [Result] Mehta SR, Tanguay JF, Eikelboom JW, Jolly SS, Joyner CD, Granger CB, Faxon DP, Rupprecht HJ, Budaj A, Avezum A, Widimsky P, Steg PG, Bassand JP, Montalescot G, Macaya C, Di Pasquale G, Niemela K, Ajani AE, White HD, Chrolavicius S, Gao P, Fox KA, Yusuf S; CURRENT-OASIS 7 trial investigators. Double-dose versus standard-dose clopidogrel and high-dose versus low-dose aspirin in individuals undergoing percutaneous coronary intervention for acute coronary syndromes (CURRENT-OASIS 7): a randomised factorial trial. Lancet. 2010 Oct 9;376(9748):1233-43. doi: 10.1016/S0140-6736(10)61088-4. PMID 20817281
- [Result] Stone GW. Acute coronary syndromes: finding meaning in OASIS 7. Lancet. 2010 Oct 9;376(9748):1203-5. doi: 10.1016/S0140-6736(10)61262-7. No abstract available. PMID 20817280
- [Derived] Bossard M, Gao P, Boden W, Steg G, Tanguay JF, Joyner C, Granger CB, Kastrati A, Faxon D, Budaj A, Pais P, Di Pasquale G, Valentin V, Flather M, Moccetti T, Yusuf S, Mehta SR. Antiplatelet therapy in patients with myocardial infarction without obstructive coronary artery disease. Heart. 2021 Nov;107(21):1739-1747. doi: 10.1136/heartjnl-2020-318045. Epub 2021 Jan 27. PMID 33504513
- [Derived] Bossard M, Granger CB, Tanguay JF, Montalescot G, Faxon DP, Jolly SS, Widimsky P, Niemela K, Steg PG, Natarajan MK, Gao P, Fox KAA, Yusuf S, Mehta SR. Double-Dose Versus Standard-Dose Clopidogrel According to Smoking Status Among Patients With Acute Coronary Syndromes Undergoing Percutaneous Coronary Intervention. J Am Heart Assoc. 2017 Nov 3;6(11):e006577. doi: 10.1161/JAHA.117.006577. PMID 29101117
- [Derived] Mehta SR, Bassand JP, Chrolavicius S, Diaz R, Fox KA, Granger CB, Jolly S, Rupprecht HJ, Widimsky P, Yusuf S; CURRENT-OASIS 7 Steering Committee. Design and rationale of CURRENT-OASIS 7: a randomized, 2 x 2 factorial trial evaluating optimal dosing strategies for clopidogrel and aspirin in patients with ST and non-ST-elevation acute coronary syndromes managed with an early invasive strategy. Am Heart J. 2008 Dec;156(6):1080-1088.e1. doi: 10.1016/j.ahj.2008.07.026. Epub 2008 Nov 1. PMID 19033002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25086 patients were enrolled and randomized between June 2006 and August 2009 in 597 sites in 39 countries. Because the observed overall blinded event rate was substantially lower than expected, the number of patients to be enrolled was increased from 18000 to 20000, then to 25000.
Pre-assignment Details: Treatment assignment was performed through an automated voice randomization service (AreS). At the same time, the AReS provided allocation to a Clopidogrel treatment regimen according to a pre-defined randomization list and to a ASA dose according to a factorial design.
Groups:
- Clopidogrel 300/75/75 mg + ASA Low Dose: Day 1: Clopidogrel 300 mg loading dose + ASA ≥ 300 mg
  Day 2 to Day 7: Clopidogrel 75 mg + ASA 75-100 mg
  Day 8 to Day 30: Clopidogrel 75 mg + ASA 75-100 mg
- Clopidogrel 300/75/75 mg + ASA High Dose: Day 1: Clopidogrel 300 mg loading dose + ASA ≥ 300 mg
  Day 2 to Day 7: Clopidogrel 75 mg + ASA 300-325 mg
  Day 8 to Day 30: Clopidogrel 75 mg + ASA 300-325 mg
- Clopidogrel 600/150/75 mg + ASA Low Dose: Day 1: Clopidogrel 600 mg loading dose + ASA ≥ 300 mg
  Day 2 to Day 7: Clopidogrel 150 mg + ASA 75-100 mg
  Day 8 to Day 30: Clopidogrel 75 mg + ASA 75-100 mg
- Clopidogrel 600/150/75 mg + ASA High Dose: Day 1: Clopidogrel 600 mg loading dose + ASA ≥ 300 mg
  Day 2 to Day 7: Clopidogrel 150 mg + ASA 300-325 mg
  Day 8 to Day 30: Clopidogrel 75 mg + ASA 300-325 mg
Period: Overall Study
Arm/Group | Clopidogrel 300/75/75 mg + ASA Low Dose | Clopidogrel 300/75/75 mg + ASA High Dose | Clopidogrel 600/150/75 mg + ASA Low Dose | Clopidogrel 600/150/75 mg + ASA High Dose
Started | 6312 (Randomized) | 6254 (Randomized) | 6267 (Randomized) | 6253 (Randomized)
TREATED WITH CLOPIDOGREL | 6271 | 6218 | 6228 | 6217
TREATED WITH ASA | 6302 | 6251 | 6261 | 6247
Completed | 6154 (Completed 30 days follow-up period) | 6107 (Completed 30 days follow-up period) | 6108 (Completed 30 days follow-up period) | 6122 (Completed 30 days follow-up period)
Not Completed | 158 | 147 | 159 | 131
Not completed — Death | 156 | 144 | 158 | 129
Not completed — Lost to Follow-up | 2 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel 300/75/75 mg + ASA Low Dose | Clopidogrel 300/75/75 mg + ASA High Dose | Clopidogrel 600/150/75 mg + ASA Low Dose | Clopidogrel 600/150/75 mg + ASA High Dose | Total
Number analyzed (Participants) | 6312 | 6254 | 6267 | 6253 | 25086
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.7) | 61.5 (11.7) | 61.2 (11.8) | 61.4 (11.9) | 61.3 (11.8)
Age, Customized [Number; unit: participants]
  < 65 years | 3792 | 3740 | 3787 | 3735 | 15054
  65 - 74 years | 1573 | 1576 | 1543 | 1543 | 6235
  ≥ 75 years | 947 | 937 | 937 | 975 | 3796
  Missing | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1702 | 1756 | 1671 | 1742 | 6871
  Male | 4610 | 4498 | 4596 | 4511 | 18215
Region of Enrollment [Number; unit: participants]
  Argentina | 182 | 159 | 162 | 174 | 677
  Australia | 97 | 100 | 96 | 95 | 388
  Austria | 41 | 35 | 35 | 40 | 151
  Belgium | 55 | 61 | 59 | 53 | 228
  Brazil | 292 | 275 | 270 | 288 | 1125
  Bulgaria | 111 | 122 | 125 | 112 | 470
  Canada | 349 | 379 | 373 | 347 | 1448
  Chile | 95 | 85 | 82 | 90 | 352
  China | 510 | 492 | 500 | 515 | 2017
  Croatia | 114 | 145 | 144 | 114 | 517
  Czech Republic | 257 | 275 | 277 | 258 | 1067
  Estonia | 1 | 0 | 0 | 1 | 2
  Finland | 132 | 127 | 127 | 132 | 518
  France | 177 | 163 | 165 | 175 | 680
  Germany | 471 | 450 | 453 | 470 | 1844
  Greece | 20 | 21 | 23 | 21 | 85
  India | 658 | 650 | 645 | 646 | 2599
  Ireland | 24 | 13 | 15 | 23 | 75
  Israel | 286 | 272 | 275 | 282 | 1115
  Italy | 232 | 260 | 258 | 231 | 981
  Korea, Republic of | 161 | 149 | 152 | 165 | 627
  Latvia | 16 | 16 | 15 | 15 | 62
  Lithuania | 26 | 31 | 30 | 28 | 115
  Malaysia | 29 | 39 | 39 | 28 | 135
  Mexico | 16 | 17 | 19 | 17 | 69
  Netherlands | 46 | 48 | 48 | 46 | 188
  New Zealand | 36 | 31 | 29 | 29 | 125
  Poland | 365 | 322 | 325 | 362 | 1374
  Romania | 47 | 30 | 33 | 48 | 158
  Russian Federation | 132 | 137 | 138 | 131 | 538
  Singapore | 10 | 13 | 15 | 10 | 48
  Slovakia | 93 | 84 | 83 | 92 | 352
  South Africa | 24 | 14 | 14 | 23 | 75
  Spain | 264 | 276 | 283 | 263 | 1086
  Sweden | 10 | 11 | 9 | 10 | 40
  Switzerland | 51 | 64 | 64 | 48 | 227
  Turkey | 79 | 96 | 94 | 78 | 347
  United Kingdom | 28 | 29 | 34 | 28 | 119
  United States | 775 | 763 | 759 | 765 | 3062
Qualifying condition [Number; unit: participants]
  Suspected Unstable Angina (UA) | 1809 | 1771 | 1757 | 1877 | 7214
  Suspected MI without ST elevation (NSTEMI) | 2662 | 2662 | 2668 | 2539 | 10531
  MI with ST elevation (STEMI) | 1839 | 1817 | 1839 | 1832 | 7327
  Missing | 2 | 4 | 3 | 5 | 14
Intended PCI performed [Number; unit: participants] — The intent to perform a PCI as early as possible and no later than 72 hours of randomization was part of the criteria for inclusion
  participants
    Yes | 4377 | 4326 | 4262 | 4298 | 17263
    No | 1935 | 1928 | 2005 | 1955 | 7823

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of CV Death / MI / Stroke - Clopidogrel Treatment Regimen Comparison
Description: The primary endpoint is the first occurrence of any of the following events:
  * Cardiovascular death (any death with a clear cardiovascular or unknown cause),
  * Myocardial Infarction (diagnosis of new Myocardial Infarction (MI) - nonfatal or fatal)
  * Stroke (presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting more than 24 hours - nonfatal or fatal)
  reported between the randomization and Day 30 (inclusive), and validated by the blinded Event Adjudication Committee (EAC).
Time Frame: 30 days
Population: The analysis is on the intent-to-treat population (ITT) that consists of all patients randomized irrespective of whether they received study medication, underwent a PCI, or otherwise complied with the study protocol.
Measure: Number; unit: participants
Groups:
- Clopidogrel 300/75/75 mg + ASA: Patients randomized to the Clopidogrel 300/75/75 mg dose regimen irrespective of the ASA dose
- Clopidogrel 600/150/75 mg + ASA: Patients randomized to the Clopidogrel 600/150/75 mg dose regimen irrespective of the ASA dose
Arm/Group | Clopidogrel 300/75/75 mg + ASA | Clopidogrel 600/150/75 mg + ASA
Number analyzed (Participants) | 12566 | 12520
participants
  CV death/MI/Stroke | 557 | 522
  - CV death | 222 | 226
  - MI (fatal or not) | 274 | 237
  - Stroke (fatal or not) | 61 | 59
Statistical Analysis 1: Comparison: Clopidogrel 300/75/75 mg + ASA vs Clopidogrel 600/150/75 mg + ASA; Test type: Superiority or Other; p = 0.3037, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by ASA dose level (low or high) and qualifying condition (UA/NSTEMI or STEMI) log-rank test; Relative Risk Reduction (%) = 6.1, 95% CI 2-sided [-5.8 to 16.6] — The relative risk reduction (high dose treatment regimen (600/150/75 mg) versus standard treatment regimen (300/75/75 mg)) is estimated using stratified Cox proportional hazards model controlling for ASA dose level and qualifying condition

2. Secondary Outcome: Occurrence of Major Bleeding - Clopidogrel Dose Regimen Comparison
Description: Major bleeding is defined as any severe bleeding (associated with any of the following: death, leading to a drop in hemoglobin ≥ 5 g/dl, significant hypotension with the need for inotropic agents, symptomatic intracranial hemorrhage, requirement for surgery or for a transfusion ≥ 4 units of red blood cells or equivalent whole blood) and other major bleeding (significantly disabling bleeding, or intraocular bleeding leading to significant loss of vision or bleeding requiring transfusion of 2-3 units of red blood cells or equivalent whole blood) after validation by the independent EAC.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Clopidogrel 300/75/75 mg + ASA | Clopidogrel 600/150/75 mg + ASA
Number analyzed (Participants) | 12566 | 12520
participants
  Major bleeding | 255 | 313
  - Severe bleeding | 195 | 236
  - Major but not severe bleeding | 65 | 83
Statistical Analysis 1: Comparison: Clopidogrel 300/75/75 mg + ASA vs Clopidogrel 600/150/75 mg + ASA; Test type: Superiority or Other; p = 0.012, Regression, Logistic — The a priori threshold for statistical significance is ≤0.05; logistic regression model including terms for ASA dose level (low or high) and qualifying condition (UA/NSTEMI or STEMI)

3. Primary Outcome: First Occurrence of CV Death / MI / Stroke - ASA Dose Comparison
Time Frame: 30 days
Population: The analysis is on the the ASA treated population that consists of all patients randomized and having receiving at least one dose of ASA. All patients were included in the treatment group to which they were allocated by the AReS.
Measure: Number; unit: participants
Groups:
- Clopidogrel + ASA Low Dose: Patients treated with ASA low dose irrespective of the Clopidogrel treatment regimen
- Clopidogrel + ASA High Dose: Patients treated with ASA high dose irrespective of the Clopidogrel treatment regimen
Arm/Group | Clopidogrel + ASA Low Dose | Clopidogrel + ASA High Dose
Number analyzed (Participants) | 12563 | 12498
participants
  CV death/MI/Stroke | 546 | 527
  - CV death | 231 | 211
  - MI (fatal or not) | 260 | 251
  - Stroke (fatal or not) | 55 | 65
Statistical Analysis 1: Comparison: Clopidogrel + ASA Low Dose vs Clopidogrel + ASA High Dose; Test type: Superiority or Other; p = 0.6047, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by clopidogrel treatment regimen (300/75/75 mg or 600/150/75 mg) log-rank test; Relative Risk Reduction (%) = 3.1, 95% CI 2-sided [-9.2 to 14.0] — The relative risk reduction (ASA high dose versus ASA low dose) is estimated using stratified Cox proportional hazards model controlling for Clopidogrel treatment regimen

4. Primary Outcome: First Occurrence of CV Death / MI / Stroke - Interaction Clopidogrel Treatment Regimen and ASA Dose Level
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Clopidogrel 300/75/75 mg + ASA Low Dose | Clopidogrel 300/75/75 mg + ASA High Dose | Clopidogrel 600/150/75 mg + ASA Low Dose | Clopidogrel 600/150/75 mg + ASA High Dose
Number analyzed (Participants) | 6312 | 6254 | 6267 | 6253
participants | 267 | 290 | 282 | 240
Statistical Analysis 1: Comparison: Clopidogrel 300/75/75 mg + ASA Low Dose vs Clopidogrel 600/150/75 mg + ASA Low Dose; Test type: Superiority or Other; p = 0.4579, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by qualifying condition (UA/NSTEMI or STEMI) log-rank test; Relative Risk Reduction (%) = -6.5, 95% CI 2-sided [-26.0 to 9.9] — The relative risk reduction (high dose treatment regimen (600/150/75 mg) versus standard treatment regimen (300/75/75 mg)) is estimated using a stratified Cox proportional hazards model controlling for qualifying condition
Statistical Analysis 2: Comparison: Clopidogrel 300/75/75 mg + ASA High Dose vs Clopidogrel 600/150/75 mg + ASA High Dose; Test type: Superiority or Other; p = 0.0262, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by qualifying condition (UA/NSTEMI or STEMI) log-rank test; Relative Risk Reduction (%) = 17.6, 95% CI 2-sided [2.2 to 30.5] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Clopidogrel 300/75/75 mg + ASA Low Dose vs Clopidogrel 300/75/75 mg + ASA High Dose vs Clopidogrel 600/150/75 mg + ASA Low Dose vs Clopidogrel 600/150/75 mg + ASA High Dose; Test type: Superiority or Other; p = 0.0355, Chi-squared — The a priori threshold for statistical significance is ≤0.05; Interaction chi-squared test of the Cox proportional hazards model

5. Primary Outcome: First Occurrence of CV Death / MI / Stroke - Clopidogrel Treatment Regimen Comparison in PCI Subgroup
Time Frame: 30 days
Population: The intent-to-treat (ITT) analysis is done on the randomized patients who underwent PCI during the study.
Measure: Number; unit: participants
Arm/Group | Clopidogrel 300/75/75 mg + ASA | Clopidogrel 600/150/75 mg + ASA
Number analyzed (Participants) | 8703 | 8560
participants
  CV death/MI/Stroke | 392 | 330
  - CV death | 132 | 130
  - MI (fatal or not) | 225 | 172
  - Stroke (fatal or not) | 35 | 28
Statistical Analysis 1: Comparison: Clopidogrel 300/75/75 mg + ASA vs Clopidogrel 600/150/75 mg + ASA; Test type: Superiority or Other; p = 0.0332, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by ASA dose level (low or high) and qualifying condition (UA/NSTEMI or STEMI) Log-rank test. No adjustment was made; Relative Risk Reduction (%) = 14.7, 95% CI 2-sided [1.2 to 26.3] — The relative risk reduction (high dose treatment regimen (600/150/75 mg) versus standard treatment regimen (300/75/75 mg)) is estimated using a stratified Cox proportional hazards model controlling for ASA dose level and qualifying condition

6. Secondary Outcome: Occurrence of Major Bleeding - ASA Dose Level Comparison
Time Frame: 30 days
Population: The analysis is on the treated patient population that consists of all patients randomized and having receiving at least one dose of ASA. All patients were included in the treatment group to which they were allocated by the AReS.
Measure: Number; unit: participants
Arm/Group | Clopidogrel + ASA Low Dose | Clopidogrel + ASA High Dose
Number analyzed (Participants) | 12563 | 12498
participants
  Major bleeding | 285 | 282
  - Severe bleeding | 215 | 216
  - Major but not severe bleeding | 74 | 73
Statistical Analysis 1: Comparison: Clopidogrel + ASA Low Dose vs Clopidogrel + ASA High Dose; Test type: Superiority or Other; p = 0.945, Regression, Logistic — The a priori threshold for statistical significance is ≤0.05; Logistic regression model including a term for Clopidogrel treatment regimen (300/75/75 mg or 600/150/75 mg)

7. Post Hoc Outcome: Occurrence of Stent Thrombosis - Clopidogrel Treatment Regimen Comparison
Description: This includes definite stent thrombosis (confirmed by angiography or evidence of recent thrombus determined at autopsy or by examination of tissue retrieved following thrombectomy) and probable stent thrombosis (unexplained death having occurred after intracoronary stenting or, MI related to acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any obvious cause) after validation by the EAC.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Clopidogrel 300/75/75 mg + ASA | Clopidogrel 600/150/75 mg + ASA
Number analyzed (Participants) | 12566 | 12520
participants
  Stent trombosis | 200 | 135
  - Definite | 111 | 58
  - Probable | 89 | 77
Statistical Analysis 1: Comparison: Clopidogrel 300/75/75 mg + ASA vs Clopidogrel 600/150/75 mg + ASA; Test type: Superiority or Other; p = 0.0004, Log Rank — The a priori threshold for statistical significance is ≤0.05; Two-sided stratified by ASA dose level (low or high) and qualifying condition (UA/NSTEMI or STEMI) log-rank test; Relative Risk Reduction (%) = 32.6, 95% CI 2-sided [16.2 to 45.8] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The analysis is on the intent-to-treat population (ITT). All patients were included in the treatment arm to which they were allocated by the AReS.
  Any adverse event that developed or worsened on or after randomization up to the day of the final follow-up visit was included.
Arm/Group | Clopidogrel 300/75/75 mg + ASA Low Dose | Clopidogrel 300/75/75 mg + ASA High Dose | Clopidogrel 600/150/75 mg + ASA Low Dose | Clopidogrel 600/150/75 mg + ASA High Dose
Serious Adverse Events (participants affected / at risk) | 322/6312 | 329/6254 | 372/6267 | 332/6253
Other Adverse Events (participants affected / at risk) | 0/6312 | 0/6254 | 0/6267 | 0/6253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel 300/75/75 mg + ASA Low Dose (N=6312) | Clopidogrel 300/75/75 mg + ASA High Dose (N=6254) | Clopidogrel 600/150/75 mg + ASA Low Dose (N=6267) | Clopidogrel 600/150/75 mg + ASA High Dose (N=6253)
Operative haemorrhage (Injury, poisoning and procedural complications) | 39 | 50 | 57 | 48
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 7 | 8 | 7 | 9
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 12 | 16 | 18 | 6
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fat embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Agitation postoperative (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Complication of device removal (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 12 | 15 | 15
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 4 | 9 | 8
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 6 | 3 | 6
Gastritis (Gastrointestinal disorders) | 2 | 3 | 2 | 3
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 4 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 21 | 11 | 22 | 16
Septic shock (Infections and infestations) | 4 | 2 | 5 | 4
Urinary tract infection (Infections and infestations) | 3 | 0 | 3 | 3
Postoperative wound infection (Infections and infestations) | 3 | 3 | 2 | 3
Bronchopneumonia (Infections and infestations) | 0 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 2 | 2 | 1 | 2
Gastroenteritis (Infections and infestations) | 4 | 1 | 1 | 2
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 2 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1
Lung infection (Infections and infestations) | 2 | 1 | 1 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 1 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1
Graft infection (Infections and infestations) | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 3 | 5 | 0
Wound infection (Infections and infestations) | 1 | 4 | 3 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 1 | 0
Application site infection (Infections and infestations) | 0 | 0 | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 3 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Catheter sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis coxsackie viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Myocarditis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Peridiverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0
Puncture site infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 17 | 21 | 22 | 31
Pyrexia (General disorders) | 1 | 5 | 0 | 4
Vessel puncture site haematoma (General disorders) | 2 | 2 | 1 | 2
Chest pain (General disorders) | 2 | 3 | 5 | 1
Multi-organ failure (General disorders) | 1 | 2 | 3 | 1
Non-cardiac chest pain (General disorders) | 4 | 2 | 2 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1
Implant site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1
Necrosis (General disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0
Application site erosion (General disorders) | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0
Mechanical complication of implant (General disorders) | 0 | 1 | 0 | 0
Implant site haematoma (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 5 | 10
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 11 | 9 | 18 | 10
Renal failure (Renal and urinary disorders) | 7 | 7 | 8 | 8
Haematuria (Renal and urinary disorders) | 5 | 4 | 4 | 5
Renal failure chronic (Renal and urinary disorders) | 2 | 2 | 0 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 2 | 2 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pericardial haemorrhage (Cardiac disorders) | 15 | 12 | 18 | 11
Intracardiac thrombus (Cardiac disorders) | 1 | 2 | 1 | 5
Pericarditis (Cardiac disorders) | 3 | 1 | 2 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac perforation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Interventricular septum rupture (Cardiac disorders) | 0 | 0 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Haemorrhage coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 6 | 7
Haemorrhage (Vascular disorders) | 3 | 5 | 5 | 2
Hypotension (Vascular disorders) | 3 | 0 | 2 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 2 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 2 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 3 | 1 | 0
Aortic dissection (Vascular disorders) | 2 | 1 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Artery dissection (Vascular disorders) | 1 | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Arterial rupture (Vascular disorders) | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Wound haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Femoral artery dissection (Vascular disorders) | 2 | 0 | 0 | 0
Venous haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 7 | 5 | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 1 | 3 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 1
Critical illness polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Drop attacks (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalomalacia (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Brain stem syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine without aura (Nervous system disorders) | 0 | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Anoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hydraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 4 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 5 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 0 | 1 | 3
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar i disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Pituitary cyst (Endocrine disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study is made jointly in the name of all wholehearted collaborators. Other papers are authored based on the contributions of the individuals to the overall study. Sub-studies with scientific merit which have received prior approvals of the Steering Committee may be published separately in the names of contributing Investigators. A copy of all manuscripts are provided to the Sponsors for their review and the final decision to publish is made by the Steering Committee.